CLINICAL TRIAL: NCT01651676
Title: Evaluation of the VQ11 Auto-questionnaire of Quality of Life in Pneumology Investigation, During the Implementation of a Long-acting Bronchodilator Treatment of Patients With COPD.
Brief Title: Estimation of the VQ11 Auto-questionnaire, to Follow Patients With Chronic Obstructive Pulmonary Disease
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PI2011_843_0006; 2011-A01653-38 (Other: ID-RCB)
Record Dates: First submitted 2012-06-29; First posted 2012-07-27 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: COPD
Keywords: VQ11 questionnaire; COPD; LBD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- COPD arm (Experimental): VQ11 validation:
  Stage II, III or IV COPD patients justifying a LABD will benefit from the studied VQ11 questionnaire
  Interventions: Other: VQ11 validation

INTERVENTIONS:
Other: VQ11 validation — Two visits per patient are planned: V1 and V2.
  For each visit, the pulmonologists ask the patients participating in the study to fill out the VQ11 questionnaire, which will be correlated to the other parameters (Likert scale, IPAQ, RFE, SGRQ,...)
  LABD treatment consist in β 2 agonists or anticholinergic drug.

SUMMARY:
The purpose of this study is to estimate the capacity of the auto-questionnaire of quality of life, VQ11, to follow the evolution of patients with COPD (Chronic obstructive pulmonary disease) in stable state (without exacerbation in the previous 6 weeks) (3 months +/-15 days) during the implementation of a LABD (Long-acting bronchodilator) treatment.

The main objective is to compare the total Score of the VQ11 auto-questionnaire before and after LABD. A decrease of 5 points of the total score mimicking an improvement in the quality of life linked to health, specifically in the COPD.

DETAILED DESCRIPTION:
Evaluation of the VQ11 auto-questionnaire of quality of life in pneumology investigation, during the implementation of a long-acting bronchodilator treatment of patients with COPD.

Two visits per patient are planned:

V1: After complete information and collection of the written consent, the pulmonologists ask the patients participating in the study to fill out the VQ11 questionnaire, 2 visual analogical scales concerning the dyspnoea and the physical activity, the short IPAQ version and the respiratory questionnaire of the Saint Georges hospital. RFE (respiratory functional exploration) is also realized during this medical exam.

V2 (3 months after the treatment setup, at day90 ± 15): the pulmonologists ask the patients participating in the study to fill out the VQ11 questionnaire, 2 visual analogical scales and Likert scales concerning the dyspnoea and the physical activity, the short IPAQ version and the respiratory questionnaire of the Saint Georges hospital. RFE (respiratory functional exploration) is also realized during this medical exam.

Inclusion period : 6 months; Study participation period / patient : 3 months; Complete study duration : 9 months

ELIGIBILITY:
Inclusion Criteria:

* COPD patient with stage II, III ou IV justifying a LABD
* Patient in stable state (without exacerbation in the previous 6 weeks)
* Clinical criteria: dyspnoea stage I ou more (MMRC scale)
* Adult over 18 years old.
* Patients naïve from LABD treatment.

Exclusion Criteria:

* Other associated pathology (bronchiectasia...)
* Heart disorder with a prevailing role in the dyspnoea
* Cardiac decompensation in the previous year
* Pregnancy and lactating
* Women in genital activity without efficient contraception method (IUD or estrogen-progestin pill)
* Lack of social insurance
* Patient non compliant to protocol, at the investigator's appreciation
* Simultaneous participation to other clinical trial.
* adult under judicial protection (tutor or curator).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
VQ11 score | V1 (at baseline), V2 (3 months after V1)
  To compare changes of total Score of the VQ11 auto-questionnaire before and after LABD (decrease of 5 points of the total score mimicking an improvement in the quality of life linked to health, specifically in the COPD).

SECONDARY OUTCOMES:
VQ11 and visual analogical scale regarding daily activity | V1 (at baseline), V2 (3 months after V1)
  To estimate the daily activity by a dedicated visual analogical scale. Variations between the two visits will be analysed in correlation to VQ11 changes.
RFE | V1 (at baseline), V2 (3 months after V1)
  Respiratory functional exploration (RFE) performed at rest (plethysmography) before and three months after LABD treatment initiation.
VQ11 sub-scores | V1 (at baseline), V2 (3 months after V1)
  To estimate the impact of an LABD treatment on patients with COPD before and three months after treatment initiation through the three sub-dimensions of the VQ11 questionnaire
Likert scales | V2 (3 months after V1)
  To estimate the evolution of dyspnoea and the daily activity by Likert scale.
VQ11 and visual analogical scales regarding dyspnoea | V1 (at baseline), V2 (3 months after V1)
  To estimate the dyspnoea by a dedicated visual analogical scale. Variations between the two visits will be analysed in correlation to VQ11 changes.
Bi-directional visual analogical scale regarding dyspnoea | V2 (3 months after V1)
  To estimate the evolution of dyspnoea since the LABD initiation.
Bi-directional visual analogical scale regarding daily activity | V2 (3 months after V1)
  To estimate the evolution of daily activity since the LABD initiation.
Saint George's Respiratory Questionnaire | V1 (at baseline), V2 (3 months after V1)
  To estimate the impact of an LABD treatment on patients with COPD before and three months after treatment initiation using the SGRQ change between the two visits.
Dyspnoea evolution assessed by mMRC | V1 (at baseline), V2 (3 months after V1)
  To estimate the impact of the LABD treatment on dyspnoea of patients with COPD before and three months after treatment initiation through the change of the Modified Medical Research Council dyspnoea scale (mMRC).

CONTACTS AND LOCATIONS:
Overall Officials: Charles DAYEN, MD, Principal Investigator — University Hospital of Amiens
Locations (17):
- France (17):
  - Clinique de l'Europe, Amiens
  - CHU Amiens Nord, Amiens
  - CHU Amiens Sud, Amiens
  - Centre Hospitalier de Chauny, Chauny
  - Centre Hospitalier de Compiègne, Compiègne
  - Centre Médical, Compiègne
  - CH Creil, Creil
  - Centre Médical, Denain
  - CH de DOUAI, Douai
  - Hopital Jacques MONOD, Le Havre
  - Centre Médical, Le Havre
  - CHRU de Lille, Lille
  - Hopital Maison Blanche, Reims
  - CHU de Rouen, Rouen
  - Centre hospitalier de St Quentin, Saint-Quentin
  - Zac Gouraud, Soissons
  - Résidence Saint Michel, Valenciennes

REFERENCES:
- [Result] https://doi.org/10.1016/j.rmr.2015.10.647 Évaluation par auto-questionnaire de qualité de vie VQ11 de l'impact d'un traitement bronchodilatateur dans la BPCO en pratique pneumologique Revue des Maladies Respiratoires Volume 33, Supplement, January 2016, Page A34